CLINICAL TRIAL: NCT06594835
Title: Pilot Test of the Better Together Intervention
Brief Title: Test of the Better Together Intervention
Acronym: BT Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00025611
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Substance Use
Keywords: substance use; feasibility; adolescents
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Better Together (Experimental): Better Together (BT) is a 90-min, an age-appropriate, culturally relevant prevention intervention to prevent substance use among Black youth experiencing household challenges (ages 11-13) by addressing the multilevel influences of substance use.
  Interventions: Behavioral: Better Together
- Control (Active Comparator): Control group participants received a media education program
  Interventions: Behavioral: Youth In the Media (YM)

INTERVENTIONS:
Behavioral: Better Together — Better Together (BT) is a 90-min, age-appropriate, culturally relevant prevention intervention to prevent substance use among Black youth experiencing household challenges (ages 11-13) by addressing the multilevel influences of substance use.
  Arms: Better Together
Behavioral: Youth In the Media (YM) — Delivered in eight in-person, 90-minute sessions concurrently with BT sessions, the YM program was designed to (1) increase participants' awareness of and access to the different types of media and free resources available at the participants local libraries, (2) discuss different types of media that center stories and experiences of Black youth, and (3) expose participants to careers in media.
  Arms: Control

SUMMARY:
Better Together (BT) is a novel, culturally relevant library-based intervention designed to prevent substance use among Black youth (ages 11-13) affected by household challenges (i.e., parental substance use, parental incarceration, and parental mental health challenges). In partnership with public and school librarians, the investigators will conduct a randomized pilot study of BT with up to 100 youth across four sites in Baltimore, Maryland to assess:

1. Implementation fidelity via logs, assessments, and observations of participants and facilitators
2. Feasibility of all key research aspects, including recruitment, randomization, intervention, and control conditions, as well as pre, post, and one-month follow-up assessments
3. Initial effects of BT on substance use

DETAILED DESCRIPTION:
This study occurred from September 2023 through May 2024 in Baltimore, Maryland, USA. The investigators partnered with two schools to assess the feasibility and acceptability of the BT intervention in a small, randomized trial. The investigators compared the outcomes of Black youth (ages 11-13) exposed to household challenges who received the intervention (n = 32) with a time-matched control group of youth exposed to household challenges (n = 27). An online random number generator was used to randomize participants to either the control or intervention group. Randomization occurred at the family level, which allowed all eligible youth from a single family to be in the same condition and minimized the potential for contamination of intervention effects. Participants completed electronic assessments three times: baseline (one week before the start of the intervention), post-test (one week after the intervention), and a 1-month follow-up (one month after the post-test). The trial ended after implementation in two schools at the end of the school year. The investigators obtained approval from the Johns Hopkins Bloomberg School of Public Health Institutional Review Board.

Youth enrollment occurred one month before the start of the intervention. To be eligible, participants had to be between 11 and 13 years old, identify as Black or African American, and have been exposed to one or more household challenges. Direct youth recruitment occurred with study team members inviting families to participate via presentations at each organization. Participants were also recruited indirectly through referrals from organizational staff and enrolled participants. Recruitment materials and presentations did not include information about household challenges as an eligibility criterion to prevent the risk of stigma associated with participating.

Interested youth were required to complete a participant interest form that included their name, as well as their caregiver's name and contact information. A study team member contacted the caregiver to inform them of the study and assist the caregiver in completing a screener to determine the youth's eligibility. A study team member reviewed the purpose and procedures of the study as outlined on the parental permission form. The permission form was emailed and texted to caregivers via Qualtrics to obtain signatures. Once permission was granted, all eligible youth in the family were assigned a participant ID. Oral assent was obtained from all youth before they completed the baseline survey.

Both intervention and control group sessions occurred twice a week, in person, during non-school hours for four weeks. At most, 15 youth were allowed to participate in each group. Sessions were co-facilitated by two study team members. Participants were compensated $25 for each session they attended and each assessment they completed.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible, participants had to be between 11 and 13 years old,
* identify as Black or African American,
* have been exposed to one or more household challenges (i.e., parental substance use, incarceration or mental illness)

Exclusion Criteria:

* Youth in foster care

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Number of Youth Retained in the intervention | From enrollment to the completion of the one-month follow-up assessment
  Retention was evaluated in two ways. First, investigators assessed retention by the number of sessions the participant attended (dosage). Investigators defined dosage success as youth participating in five or more sessions. Second, retention was assessed by the proportion of youth who completed the post-test and 1-month follow-up. Investigators defined retention success as more than 80% of the sample was retained at all assessments.

SECONDARY OUTCOMES:
Number of Youth who use any substance | From baseline to one-month follow-up
  One item was used to assess substance use behaviors: "Have you ever had a drink of alcohol (more than a few sips) or tried any drug (i.e., marijuana, cigarette, prescription pills, ecstasy, cocaine, etc.)?" Participants responded, 'yes' or 'no'.
Substance use knowledge as assessed by survey | From baseline to one-month follow up
  Three true/false items were used to assess substance use knowledge: (1) alcohol is considered a drug, (2) drinking alcohol or using drugs leads to poor judgment and decision-making, and (3) it is against the law for children and teenagers to use drugs. Correct responses were summed to create a scale ranging from 0 to 3. with higher scores indicating more knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Terrinieka Powell, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Powell TW, Offiong A, Lewis Q, Prioleau M, Smith B, Johnson RM. "I've smoked weed with my daughter": Cannabis Use within Families Affected by Parental Opioid Misuse. Child Youth Serv Rev. 2023 Dec;155:107235. doi: 10.1016/j.childyouth.2023.107235. Epub 2023 Oct 15. PMID 37982095
- See also: Website for the research team — https://www.researchbypowell.com